CLINICAL TRIAL: NCT04716699
Title: Assessing Systemic and Local Levels of Lidocaine During Surgery for Glioblastoma
Brief Title: Systemic and Local Levels of Lidocaine During Surgery for the Removal of Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kiarash Shahlaie, M.D., Ph.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Kiarash Shahlaie, M.D., Ph.D., Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UCDCC#285; NCI-2020-14099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#285 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (lidocaine, surgery) (Experimental): Patients receive bolus lidocaine IV per standard of care. After intubation, patients receive another infusion of lidocaine IV over 4 hours or until the end of surgery. Patients also undergo collection of blood and tumor samples at the start of surgery and hourly afterwards until a total of 4 samples are collected.
  Interventions: Procedure: Biospecimen Collection; Drug: Lidocaine; Procedure: Resection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tumor samples
Drug: Lidocaine — Given IV
  Other Names: .omega.-Diethylamino-2,6-dimethylacetanilide; 2-(Diethylamino)-2'',6''-acetoxylidide; Cuivasil; Duncaine; Leostesin; Lidothesin; Lignocaine; Rucaina
Procedure: Resection — Undergo surgical resection per standard of care
  Other Names: Surgical Resection

SUMMARY:
This clinical trial measures the amount and effect of lidocaine injected into patients with glioblastoma while they are undergoing surgical removal of their brain tumors. Lidocaine is a substance used to relieve pain by blocking signals at the nerve endings in skin. Information gained from this study may help researchers come up with new treatments to help patients with glioblastomas in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the pharmacokinetic properties of intravenously administered lidocaine inside a glioblastoma tumor by means of mass spectroscopy.

SECONDARY OBJECTIVE:

I. To assess the differences in overall survival (OS) and progression free survival (PFS) between the patients in the lidocaine therapy group and historical controls taken from the literature (Stupp et al) with comparable post-operative treatment regimen.

OUTLINE:

Patients receive bolus lidocaine intravenously (IV) per standard of care. After intubation, patients receive another infusion of lidocaine IV over 4 hours or until the end of surgery. Patients also undergo collection of blood and tumor samples at the start of surgery and hourly afterwards until a total of 4 samples are collected.

After completion of surgery, patients are followed for 24 hours, and at 7-14 days, up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Preoperative imaging characteristics consistent with brain glioblastoma (magnetic resonance imaging [MRI] brain)
* Patients who are undergoing neurosurgical resection for treatment of glioblastoma
* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Prior treatment for glioblastoma
* Glioblastoma size less than 5 cm^3
* Known allergy against amide type of local anesthetics
* History of severe cardiac failure (determined by clinical history of less the 3 Metabolic Equivalent of Tasks [METs])
* 2nd or 3rd degree heart block (exception: patients with pacemaker)
* Concurrent treatment with class I or III antiarrhythmics (phenytoin, procainamide, propranolol, quinidine) or amiodarone use =< 3 months
* History of Wolff-Parkinson-White syndrome, Stokes Adams syndrome, or active dysrhythmia
* History of bradycardia
* Prior clinical history of severe hepatic impairment or alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 1.55 times of upper normal limit
* Prior clinical history of severe renal impairment or estimated glomerular filtration rate (EGFR) < 30ml/min
* Uncontrolled seizure disorder
* Acute porphyria
* Patients requiring an awake fiberoptic intubation due to administration of additional lidocaine
* Pregnant or lactating women
* Any condition that would prohibit the understanding or rendering of informed consent
* Any medical condition including additional malignancies, laboratory abnormalities, or psychiatric illness that in the opinion of the investigator would prevent the subject from participating and adhering to study related procedures
* Uncontrolled concomitant disease that in the opinion of the investigator would interfere with the patient's safety or compliance on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-12-26 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Difference between the concentrations of lidocaine in the tumor tissue and in the blood (baseline level) | At start of surgery up until completion of surgery, assessed up to 4 hours after starting surgery
  Analysis is mainly descriptive and will be mainly done by Lidocaine analysis lab. Will report the mean and standard deviation of concentration of lidocaine in the tumor and blood at 3 time points. The pharmacokinetics of lidocaine within the tumor will be summarized using the means, and standard pharmacokinetics parameters will be reported (maximum concentration, time of maximum concentration, and area under the curve). If applicable, will use mixed effects model to summarize trajectories of change for concentration measured at multiple time points, which will account for correlation between repeated measures within patient.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From diagnosis to first documented evidence of disease progression or death, whichever comes first, assessed up to 30 days after surgery
  Kaplan-Meier plots and confidence intervals will be used to summarize PFS. Medians (and associated 95% confidence intervals) of PFS will then be calculated and compared with historical control from the literature.
Overall survival (OS) | From diagnosis to death, assessed up to 30 days after surgery
  Kaplan-Meier plots and confidence intervals will be used to summarize OS. Medians (and associated 95% confidence intervals) of OS will then be calculated and compared with historical control from the literature.
Incidence of adverse events (AEs) | Up to 30 says after surgery
  Will record safety and toxicity profile using National Cancer Institute Common Terminology Criteria for Adverse Events 5.0. AEs will be summarized using descriptive statistics. The type, grade, frequency and proportion of toxicities will be reported, along with associated 95% confidence interval of proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Kiarash Shahlaie, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States